CLINICAL TRIAL: NCT06622005
Title: Phase 1 Trial of SX-682, a CXCR 1/2 Inhibitor, in Combination With Standard of Care Treatment in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: SX-682 in Combination With Carfilzomib, Daratumumab-Hyaluronidase, and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3850824
Record Dates: First submitted 2024-09-30; First posted 2024-10-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Hyaluronoglucosaminidase; carfilzomib; Dexamethasone; Calcium Dobesilate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Patients receive SX-682 PO BID on days 1-21 of each cycle. Patients also receive daratumumab-hyaluronidase SC once weekly on cycles 1 and 2 and once every 2 weeks on cycles 3-6 and carfilzomib IV on days 1, 8 and 15 and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with sustained response after 6 cycles may continue to receive SX-682 PO BID on days 1-21, daratumumab-hyaluronidase SC on day 1, carfilzomib IV on days 1, 8, and 15 and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, BM aspiration, ECHO and PET/CT or MRI on study.
  Interventions: Drug: Cxcr1/2 Inhibitor SX-682; Drug: Daratumumab and Recombinant Human Hyaluronidase; Drug: Carfilzomib; Drug: Dexamethasone; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Echocardiography; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Cxcr1/2 Inhibitor SX-682 — Given PO
  Other Names: SX-682
Drug: Daratumumab and Recombinant Human Hyaluronidase — Given SC
  Other Names: Daratumumab and hyaluronidase
Drug: Carfilzomib — Given IV
  Other Names: CFZ; PR 171
Drug: Dexamethasone — Given PO
  Other Names: Adexone; Baycadron; Cortidexason; Decadrol; Fluorodelta; Loverine
Procedure: Biospecimen Collection — Undergo Blood sample collection
Procedure: Bone Marrow Aspiration — Undergo Bone Marrow Aspiration
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: PET; PET Scan
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI Scan

SUMMARY:
This phase I trial tests the safety and side effects of SX-682 in combination with standard of care treatment carfilzomib, daratumumab-hyaluronidase, and dexamethasone in treating patients with multiple myeloma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). SX-682 works by blocking certain sites on cells that suppress the ability of the immune system to destroy tumor cells. Blocking those specific sites allows other cells of the immune system to become "free" to kill tumor cells. Carfilzomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and tumor cells, including myeloma cells. Daratumumab may block CD38 and help the immune system kill tumor cells, while hyaluronidase helps to deliver daratumumab to CD38-expressing tumor cells through a subcutaneous injection. Dexamethasone is in a class of medications called corticosteroids. It is known to kill myeloma cells and is also used to reduce inflammation and lower the body's immune response to monoclonal antibodies like dratumumab and help lessen its side effects. Giving SX-682 in combination with carfilzomib, daratumumab-hyaluronidase and dexamethasone may be safe and tolerable in treating patients with relapsed or refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Confirmed relapsed/ refractory multiple myeloma
* Measurable disease including at least one of the following criteria:

  * Serum M-protein ≥ 0.5 g/dL
  * Urine M-protein ≥ 200 mg/24h
  * Serum free light chain assay: involved free light chain (FLC) level greater or equal to 100 mg/L provided serum free light chain ratio is abnormal
  * Bone marrow plasma cells ≥ 10% total bone marrow cells
* ≥ 1 prior line of therapy
* Planned treatment with a carfilzomib/daratumumab/dexamethasone regimen
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count: ≥ 3 x 10^9/L
* Platelets: ≥ 75 x 10^9/L
* Hemoglobin: ≥ 7 g/dL
* Total bilirubin: ≤ 1.5 x upper limit of normal (ULN): ≤ 3.0 x ULN for Gilbert's syndrome
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]): ≤ 3 x ULN
* Renal Function: Estimated creatinine clearance ≥ 45 mL/min (Cockroft-Gault)
* Left ventricular ejection fraction of at least 50%
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 6 months following the last dose of the investigational drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients with non-secretory myeloma, systemic light chain amyloidosis or, plasmacytoma
* Intolerance to SX-682 or any other of the treatment components
* Refractory to prior carfilzomib (i.e. relapse or progression on or within 60 days after completion of treatment)
* Refractory to prior daratumumab (i.e. relapse or progression on or within 60 days after completion of treatment)
* Concomitant medication(s) known to be (a) a strong inhibitor or inducer of CYP3A4, or (b) QT prolonging as defined in the drug's approved label, with the exception of drugs that are considered absolutely essential for the care of the subject or if the investigator believes that beginning therapy with such medication is vital to an individual subject's care while on study, and in either case, there is no alternative medication
* Electrocardiogram (ECG) demonstrating a corrected QT (QTc) interval > 470 msec or patients with congenital long QT syndrome
* Coronary artery bypass, angioplasty, vascular stent, myocardial infarction, angina or congestive heart failure in the last 6 months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, class III or IV heart failure (New York Heart Association functional classification system) or psychiatric illness/social situations that would limit compliance with study requirements
* History of hepatitis B, C or HIV
* Known active bacillus tuberculosis infection
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-04-10 (Estimated); Study Completion 2030-04-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | WIthin the first 28 days of start of treatment
  Dose limiting toxicities will be summarized using frequencies and relative frequencies. Estimates of the dose-limiting toxicity rates will be obtained with 90% credible regions obtained by Jeffrey's prior method. The summary will be performed by dose level, if applicable.

SECONDARY OUTCOMES:
Percentage of Overall response rate | Up to 3 years after last patient is enrollled
  Obtained using Jeffrey's prior method
Percentage of Progression-free survival | Up to 3 years after last patient is enrolled
  Determined using Kaplan-Meier estimates
Percentage of Overall Survival | Up to 3 years after last patient is enrolled
  Determined using Kaplan-Meier estimates
Incidence of Adverse Events (AE's_ | Within the first 6 months of treatment
  AE's will be grading using CTCAE v.5.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hillengass, MD, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States